CLINICAL TRIAL: NCT01371097
Title: The Effect of Progressive Resistance Strength Training in Hospitalised Elderly Patients
Brief Title: Progressive Resistance Strength Training (PRT) in Hospitalised Elderly Patients
Acronym: B15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Sigrid Tibaek, Dr Med Sci, pt, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-KA-2006-0144
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Medical Diseases; Neurological Diseases; Chronical Obstructive Lung Diseases
Keywords: Barthel Index; elderly hospitalised patients; progressive resistance training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention)
- Treatment group (Experimental)
  Interventions: Other: Progressive Resistance strength training

INTERVENTIONS:
Other: Progressive Resistance strength training — Resistance strength training is given as circle training. The resistance is increased with regularly intervals.
  Arms: Treatment group

SUMMARY:
The aim of the study is to evaluate the effect of progressive resistance strength training (PRT) in elderly hospitalised patients. The hypothesis is that PRT given as an additional training would improve the rehabilitation and increase the level of activity of daily living.

DETAILED DESCRIPTION:
Elderly inpatients included in the study were randomised into a control group or a training group. All included patients received the regular in-physiotherapy, but the training group received progressive resistance training in groups in addition.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalised elderly patients referred for physiotherapy.
2. Ability to perform standing position independently with/without walking aids (rollator, crutch) or bed/bench support.

Exclusion Criteria:

1. Expected length of stay < 7 days.
2. Dementia.
3. Unable to communicate relevant.
4. Unable to be active

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Timed "Up & Go" Test | Before randomisation and 3 days before discharge from the department
  The Timed Up & Go (TUG) test assess basic functional mobility.(14). The test measures the time (in seconds)that the subjects used for standing up from the seating position on a chair (chair seat height = 45 cm) with armrest, walking 3 m, turning around and walking back to the chair and sitting down again.

SECONDARY OUTCOMES:
Barthel Index | before randomisation and 3 days before discharge from the department
  BI consists of 10 functional tasks of which 3 tasks focus the function of mowing and walking. Task numbers 8 in BI "Transfer" assess the ability to move and are rated on a 0, 5 and10 point ordinal scale. Task number 9 in BI "Walking" assess the ability to walk rated on a 0, 5 or 10 point scale.
  Task number 10 in BI "Stairs" assesses the ability to walk on stairs and is rated with 0, 5, 10 or 15 points.

CONTACTS AND LOCATIONS:
Overall Officials: Sigrid Tibaek, Dr Med Sci, PT, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Copenhagen University Hospital, Glostrup, Glostrup Municipality, Denmark